CLINICAL TRIAL: NCT01960205
Title: Effect of Saxagliptin on Body Fat , Glucose and Beta Cell Function in Patients With Newly Diagnosed Pre-Diabetes Mellitus and Obesity
Brief Title: Effect of Saxagliptin on Pre-Diabetes Mellitus and Obesity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Collaborators: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Xinli Zhou，MD，PHD, Xinli Zhou, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZXL-201308
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Prediabetes
Keywords: Saxagliptin, prediabetes, glucose intolerance,obesity
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Obesity | interventions — saxagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standarddose Saxagliptin (Experimental): Saxagliptin 5 mg (tablet) ,5mg a day and lifestyle intervention for 6 months
  Interventions: Drug: Saxagliptin
- Lifestyle intervention (Active Comparator): Lifestyle intervention for 6 months
  Interventions: Other: lifestyle intervention
- Metformin (Active Comparator): Metformin 500 mg (tablet) ,500mg three times a day and lifestyle intervention for 6 months
  Interventions: Drug: metformin
- low dose Saxagliptin (Experimental): Saxagliptin 5 mg (tablet) ,2.5 mg a day and lifestyle intervention for 6 months
  Interventions: Drug: saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — 5mg a day for 6 months
  Other Names: Onglyza
  Arms: Standarddose Saxagliptin
Drug: saxagliptin — 2.5 mg a day for 6 months
  Other Names: Onglyza
  Arms: low dose Saxagliptin
Drug: metformin — 500mg three times a day for 6 months
  Other Names: melbine
  Arms: Metformin
Other: lifestyle intervention — lifestyle intervention for 6 months
  Other Names: living way intervention
  Arms: Lifestyle intervention

SUMMARY:
The purpose of the study is to examine the effect of Saxagliptin in the newly diagnosed people with pre-diabetes and obesity besides lifestyle intervention ,there to evaluate DPP 4 inhibitors of reversing pre-diabetes curative effect to normal blood sugar, and observe its influences on the targets of obesity related metabolic abnormalities, to explore new ways for intervention on populations with pre-diabetes and obesity .

DETAILED DESCRIPTION:
Materials and Methods: This is a perspectiveness ,randomized, opening study, patients will be randomly assigned to the standarddose Saxagliptin group ,the lifestyle intervention group,the Metformin group and the low dose Saxagliptin group with a 6-month treatment period.

Oral glucose tolerance test will examined before and 6 months post-treatment during the trial.

ELIGIBILITY:
Inclusion Criteria:

1.Newly diagnosed insulin resistance or glucose intolerance .

2.20 to 70 years of age.

3.BMI≥28kg/m2，or BMI>25kg/m2 beside waistline≥80cm（female)，≥90cm(male).

Exclusion Criteria:

1. Under Diabetes Mellitus treatment.
2. Allergy to dipeptidyl peptidase 4 (DPP-4) inhibitors .
3. Active heart failure.
4. Unwilling or unable to sign inform consents.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
oral glucose tolerance test | Change of Blood sugar from baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xinli Zhou, MD, PhD, Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

REFERENCES:
- [Derived] Wang Z, Xu D, Huang L, Zhang T, Wang J, Chen Q, Kong L, Zhou X. Effects of saxagliptin on glucose homeostasis and body composition of obese patients with newly diagnosed pre-diabetes. Diabetes Res Clin Pract. 2017 Aug;130:77-85. doi: 10.1016/j.diabres.2017.05.012. Epub 2017 May 12. PMID 28575729